CLINICAL TRIAL: NCT04812002
Title: Phase II Single-arm Clinical Study of PD-1 Antibody and Bevacizumab in the Treatment of Relapsed or Refractory High-risk Gestational Trophoblasitc Neoplasia After Second-line or Above Combined Chemotherapy
Brief Title: Study of PD-1 Antibody and Bevacizumab in the Treatment of High-risk GTN After Combined Chemotherapy
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Women's Hospital School Of Medicine Zhejiang University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CSEM018
Record Dates: First submitted 2021-03-21; First posted 2021-03-23 (Actual); Last update posted 2022-06-03 (Actual); Status verified 2022-06

CONDITIONS: Gestational Trophoblastic Neoplasia
Keywords: bevacizumab; pd-1; chemotherapy
MeSH Terms: conditions — Gestational Trophoblastic Disease; Parkinson Disease 4, Autosomal Dominant Lewy Body | interventions — camrelizumab; Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Double medicine combined (Experimental): participants received 200mg of PD-1 inhibitors combined 15mg of bevacizumab per square body surface area intravenously every 3 weeks
  Interventions: Drug: PD-1 inhibitor， bevacizumab

INTERVENTIONS:
Drug: PD-1 inhibitor， bevacizumab — Both drugs are given intravenously
  Other Names: Camrelizumab for Injection

SUMMARY:
Gestational trophoblastic Neoplasia（GTN） is a kind of malignant tumor in women of childbearing age. It is easy to metastasized through the blood system in the early stage, so it is a relatively malignant tumor. The tumor is highly sensitive to chemotherapy, and low-risk patients have good prognosis, with survival rate and cure rate approaching 100%, but high-risk patients are prone to drug resistance, or relapse after remission. For relapsed, refractory, high-risk GTN, multiple remedies have been reported in the literature, but the remission rate is only 75-80%. For relapsed or refractory high-risk GTN, multiple remedies have been reported in the literature, but the remission rate is only 75-80%.

Currently, targeted therapy and immunotherapy are widely used in various refractory solid tumors. For GTN, there are also a number of related studies. In this study, PD-1 inhibitors combined with bevacizumab were used to treat refractory high-risk GTN with relapse or drug resistance after receiving previous second-line or above multidrug combination therapy, to study the efficacy and safety of the treatment regimen.

DETAILED DESCRIPTION:
In this study, PD-1 inhibitors combined with bevacizumab were used to treat refractory high-risk trophoblastic tumor (GTN) with relapse or drug resistance after receiving previous two-line or above multidrug combination therapy, and the efficacy and safety of the two drugs were evaluated.

Patients who meet the requirements will sign the informed consent and be enrolled voluntarily. This project is a single-arm study without a control group. Twenty patients are expected to be enrolled, and there are 4 centers competing for enrollment.

All patients received at least two-line multidrug combination therapy, and some patients may have undergone or planned surgery and/or radiation therapy. Through the HCG value and measurable changes in the size of the lesions, we can understand the changes of the disease. The primary endpoints were PFS and ORR Whenever, for whatever reason, the subject does not complete the clinical trial observation, is considered to be an abscission case. When the subject falls off, the researcher must fill in the reason for the fall off in the CRF, and contact the subject as much as possible, complete the items that can be evaluated, and record the time of the last medication to prepare for the analysis of its efficacy and safety. The CRF should be kept for future reference

ELIGIBILITY:
Inclusion Criteria:

1. Signed Informed Consent
2. Clinically diagnosed as recurrent or drug-resistant trophoblastic tumor
3. After treatment with at least two or more multidrug chemotherapy regimens
4. Survival is expected to exceed 3 months
5. Age ≥18 years, age ≤75 years
6. Karnofsky score ≥60分，ECOG score ≤2分
7. No serious complications
8. Take effective contraceptives during treatment
9. Patients can be followed up as required
10. Blood test within 3 days: ANC≥1.5×109/L, PT ≥100×109/L, Hb≥90g/L, BIL ≤ 1.5 times of the high limit of normal value, ALT/ALST ≤ 1.5 times of the high limit of normal value, BUN and Cr≤ normal value
11. Coagulation function, thyroid function and myocardial enzyme in the normal range

Exclusion Criteria:

1. Previously, he had received anti-PD-1, anti-PD-L1, bevacizumab and other drugs;
2. Within 2 weeks before the first administration, he had received anticancer Chinese patent medicine or immunomodulatory drugs;
3. Within 2 years before the first administration, he had received active autoimmune disease requiring systemic treatment;
4. Were receiving systemic glucocorticoid therapy or any other form of immunosuppressive therapy within 7 days prior to first administration;
5. Clinically uncontrollable pleural effusion/peritoneal effusion is present;
6. Allergic to PD-1 monoantibody, bevacizumab and other active ingredients or excipients；
7. Failure to fully recover from toxicity and/or complications；
8. History of HIV infection, untreated active hepatitis B, and active HCV infection subjects；
9. Live vaccine was administered within 30 days prior to the first dose；
10. Patients with serious or uncontrollable medical conditions who are not suitable for chemotherapy；
11. Participating in clinical trials of other drugs at the same time or 4 weeks before the first administration。

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2021-04-15 (Actual); Primary Completion 2024-04-15 (Estimated); Study Completion 2026-04-15 (Estimated)

PRIMARY OUTCOMES:
PFS | From date of randomization until the date of first documented progression or death from any cause, whichever occurred first, or last follow-up for patients alive without progression, assessed up to approximately 24 months
  PFS is defined as the time from randomization to the first occurrence of PD, as determined by the investigator using RECIST v1.1, or death from any cause during the study, whichever occurs first.

SECONDARY OUTCOMES:
ORR | From date of randomization until PD or death from any cause, assessed up to 24 months
  ORR is defined as the rate of CR or PR.Partial response (PR) is defined as a reduction of HCG by 50% or more from the starting value in continuous measurements; Complete response (CR) is defined as HCG normalization of continuous measurements at least two weeks intervals.

CONTACTS AND LOCATIONS:
Overall Officials: Xing Xie, doctor, Principal Investigator — Women's Hospital School Of Medicine Zhejiang University
Locations (1):
- Women's Hospital School of Medicine Zhejiang University, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lurain JR, Singh DK, Schink JC. Primary treatment of metastatic high-risk gestational trophoblastic neoplasia with EMA-CO chemotherapy. J Reprod Med. 2006 Oct;51(10):767-72. PMID 17086804
- [Background] Alifrangis C, Agarwal R, Short D, Fisher RA, Sebire NJ, Harvey R, Savage PM, Seckl MJ. EMA/CO for high-risk gestational trophoblastic neoplasia: good outcomes with induction low-dose etoposide-cisplatin and genetic analysis. J Clin Oncol. 2013 Jan 10;31(2):280-6. doi: 10.1200/JCO.2012.43.1817. Epub 2012 Dec 10. PMID 23233709
- [Background] Li J, Yue H, Wang X, Chen R, Lu X. Chemotherapy for gestational trophoblastic neoplasia patients with a FIGO score of 12 or greater: A multistudy analysis. Eur J Obstet Gynecol Reprod Biol. 2019 Jul;238:164-169. doi: 10.1016/j.ejogrb.2019.05.023. Epub 2019 May 20. PMID 31136884
- [Background] Anantharaju AA, Pallavi VR, Bafna UD, Rathod PS, R VC, K S, Kundargi R. Role of salvage therapy in chemo resistant or recurrent high-risk gestational trophoblastic neoplasm. Int J Gynecol Cancer. 2019 Mar;29(3):547-553. doi: 10.1136/ijgc-2018-000050. Epub 2019 Jan 29. PMID 30700567
- [Background] Bianconi MI, Otero S, Storino C, Jankilevich G. Role of Capecitabine in the Management of Gestational Trophoblastic Neoplasia: A Drug for Two Settings. J Reprod Med. 2017 May-Jun;62(5-6):250-6. PMID 30027717
- [Background] Wang J, Short D, Sebire NJ, Lindsay I, Newlands ES, Schmid P, Savage PM, Seckl MJ. Salvage chemotherapy of relapsed or high-risk gestational trophoblastic neoplasia (GTN) with paclitaxel/cisplatin alternating with paclitaxel/etoposide (TP/TE). Ann Oncol. 2008 Sep;19(9):1578-83. doi: 10.1093/annonc/mdn181. Epub 2008 May 2. PMID 18453518
- [Background] Bolze PA, Patrier S, Massardier J, Hajri T, Abbas F, Schott AM, Allias F, Devouassoux-Shisheboran M, Freyer G, Golfier F, You B. PD-L1 Expression in Premalignant and Malignant Trophoblasts From Gestational Trophoblastic Diseases Is Ubiquitous and Independent of Clinical Outcomes. Int J Gynecol Cancer. 2017 Mar;27(3):554-561. doi: 10.1097/IGC.0000000000000892. PMID 28060141
- [Background] Veras E, Kurman RJ, Wang TL, Shih IM. PD-L1 Expression in Human Placentas and Gestational Trophoblastic Diseases. Int J Gynecol Pathol. 2017 Mar;36(2):146-153. doi: 10.1097/PGP.0000000000000305. PMID 27362903